CLINICAL TRIAL: NCT01543087
Title: A PHASE 3 STUDY TO ASSESS THE PERSISTENCE OF HSBA RESPONSE UP TO 48 MONTHS AFTER COMPLETION OF A PRIMARY SERIES OF BIVALENT RLP2086, AND THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A BOOSTER DOSE OF BIVALENT RLP2086
Brief Title: Duration of hSBA Response After a Primary Series of Bivalent rLP2086 Followed by a Booster Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Other
Other Study IDs: B1971033; 2011-005697-31 (EudraCT Number)
Record Dates: First submitted 2012-02-17; First posted 2012-03-02 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-02

CONDITIONS: Meningococcal Infection
MeSH Terms: conditions — Meningococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One group of subjects (Other)
  Interventions: Procedure: blood sampling; Drug: bivalent rLP2086

INTERVENTIONS:
Procedure: blood sampling — Blood sample collection at different time points
Drug: bivalent rLP2086 — A booster dose of bivalent rLP2086 at approximately 48 months following the final dose of the 2- or 3-dose primary bivalent rLP2086 vaccination series will be given at Visit 7.

SUMMARY:
This study is to assess the longevity of immune response in adolescents for approximately 48 months after receipt of a primary series of bivalent rLP2086 vaccination, which is then followed by a booster dose and an assessment of immune response for 12 or 26 months post booster vaccination.

DETAILED DESCRIPTION:
This study is to assess the longevity of immune responses in adolescents (aged 10 to <19 years at the time of entry into a primary study) following receipt of a vaccination regimen of 2 or 3 doses of bivalent rLP2086 in a primary study. A booster dose of bivalent rLP2086 at approximately 48 months was given following the final dose of the 2- or 3-dose primary bivalent rLP2086 vaccination series. The study was therefore divided into Stage 1 (4-year persistence of immune responses following receipt of a primary vaccination series) and the booster stage (follow-up through 12 months for all boosted or 26 months for a subset of the boosted).

Subjects participating only in Stage 1 will attend up to 6 study visits for collection of a 20-mL blood sample at each visit. Subjects participating in both Stage 1 and booster stage will attend up to 9-10 study visits with 1 visit for booster dose vaccination and 8-9 visits for collection of a 20-mL blood sample at each visit.

ELIGIBILITY:
Inclusion Criteria for Stage 1:

1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. Subjects who are willing and able to comply with scheduled visits, laboratory tests, and other study procedures.
3. Subjects who completed a primary study and received all the scheduled injections within the originally planned schedule, either with bivalent rLP2086 (either 2 or 3 doses) or with investigational product in cases where subject vaccine assignment is blinded at the time of consent for study B1971033.
4. Subjects who completed the blood draw following the last vaccination and subjects who completed the 6-month follow-up telephone call in the primary study.

Inclusion Criteria for Booster Stage Visits 7-10 (up to12 month post booster follow up):

1. Evidence of a personally signed and dated ICD indicating that the subject or subject's parent(s)/legal guardian has been informed of all pertinent aspects for Visits 7 to 10 of the booster stage of the study.
2. Subject continues to meet all Stage 1 inclusion and none of the Stage 1 exclusion criteria.
3. Subject is confirmed as having received bivalent rLP2086 in the primary vaccination study.
4. Subject has completed B1971033 Stage 1 and completed the Visit 6 blood draw.
5. Subject is available for the entire period of the booster stage and the subject or subject's parent(s)/legal guardian can be reached by telephone.
6. Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
7. Male and female subjects of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception through Visit 10 of the booster stage. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active. Refer to Section 4.5 for further information.
8. Negative urine pregnancy test for all female subjects on the day of the booster dose.

Inclusion Criteria for Booster Stage Visit11 (26 month post booster follow up):

1. For subject participating in Visit 11, evidence of a personally signed and dated ICD indicating that the subject or subject's parent(s)/legal guardian has been informed of all pertinent aspects of Visit 11.
2. Subject continues to meet all Stage 1 inclusion and none of the Stage 1 exclusion criteria.
3. Subject must have received 2 or 3 doses of bivalent rLP2086 in the primary study on a 0-, 2-, and 6-month or a 0- and 6-month schedule.
4. Subject must have completed booster vaccination at Visit 7.

Exclusion Criteria for Stage 1:

1. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the trial.
2. With the exception of the primary study of bivalent rLP2086, participation in other studies within the 1-month (30-day) period before study Visit 1 and/or during study participation. Participation in purely observational studies is permitted.
3. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
4. History of culture-proven disease caused by N meningitidis or Neisseria gonorrhoeae.
5. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate blood draw.
6. Receipt of any blood products, including gamma globulin, in the period from 6 months before any study visit.
7. Vaccination with any licensed or experimental meningococcal serogroup B vaccine since being enrolled in the primary Pfizer-sponsored MnB study (other than study vaccines permitted in the primary study).
8. Subjects who were not compliant with primary study eligibility criteria while enrolled in the primary study.

Exclusion Criteria for Booster Stage:

1. Subjects who are scheduled to receive 1 or more doses of a human papillomavirus (HPV) vaccine as part of a 3-dose series during the 28 days after the booster vaccination.
2. A previous anaphylactic reaction to any vaccine or vaccine-related component.
3. Subjects receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
4. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
5. A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B-cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects in the United States with terminal complement deficiency are excluded from participation in this study. Please refer to the study reference manual (SRM) for additional details.
6. Significant neurological disorder or history of seizure (excluding simple febrile seizure).
7. Current chronic use of systemic antibiotics.
8. Current participation in another investigational study. Participation in purely observational studies is acceptable.
9. Received any investigational vaccines, drugs, or devices within 28 days before administration of the booster vaccination.
10. Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
11. Pregnant female subjects, breastfeeding female subjects, male subjects with partners who are currently pregnant, or male and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol through Visit 10 of the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 698 (Actual)
Dates: Start 2012-09-07 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (36):
  - Clinical Research Advantage, Inc. / East Valley Family Physicians, PLC, Chandler, Arizona
  - Clinical Research Advantage, Inc./ East Valley Family Physicians, PLC, Chandler, Arizona
  - St. Joseph Heritage Healthcare, Huntington Beach, California
  - Center For Clinical Trials, LLC, Paramount, California
  - California Research Foundation, San Diego, California
  - Bayview Research Group, Valley Village, California
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - USF Health, Tampa, Florida
  - North Georgia Research Clinical Center, Dalton, Georgia
  - Pediatrics and Adolescent Medicine, PA, Marietta, Georgia
  - Pediatrics And Adolescent Medicine, P.A., Woodstock, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Clinical Research Advantage, Inc., Council Bluffs, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - U of L Pediatrics: Downtown, Louisville, Kentucky
  - Brownsboro Park Pediatrics, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Southwestern Medical Clinic Lakeland Healthcare Affiliate, Stevensville, Michigan
  - The Center For Pharmaceutical Research, Kansas City, Missouri
  - Clinical Research Advantage, Inc. (Prairie Fields Family Medicine, PC), Fremont, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Creighton University Pediatric Infectious Diseases, Omaha, Nebraska
  - Clinical Research Center of Nevada,LLC, Henderson, Nevada
  - Dr. Shelly David Senders MD Inc. dba Senders Pediatrics, Cleveland, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Ohio Pediatrics, Inc, Dayton, Ohio
  - West Houston Clinical Research Service (WHCRS), Houston, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - BB Holdings, LLC., dba Jean Brown Research, Salt Lake City, Utah
  - J. Lewis Research Inc, Jordan River Family Medicine, South Jordan, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - The Vancouver Clinic, Inc. PS, Vancouver, Washington
  - Monroe Clinic, Monroe, Wisconsin
  - Research and Education Association for Clinical Health, Inc., Monroe, Wisconsin
- Czechia (9):
  - Ordinace praktickeho lekare pro deti a dorost, Holice
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Ordinace praktickeho lekare pro deti a dorost, Odolena Voda
  - Ordinace praktickeho lekare pro deti a dorost, Pardubice
  - Ordinace praktickeho lekare pro deti a dorost, Prague
  - Ordinace praktickeho lekare pro deti a dorost, Praha - Nusle
  - Ordinace praktickeho lekare pro deti a dorost, Sezemice
- Aarhus University hospital Skejby, Aarhus N, Denmark
- Finland (4):
  - Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - Pori Vaccine Research Clinic, Pori
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- Germany (2):
  - Kinder - und Jugendarzt Praxis, Bad Saulgau
  - Kinderarzt Praxis, Bramsche
- Sweden (2):
  - Infektionskliniken Malarsjukhuset, Eskilstuna
  - Skanes Universitetssjukhus, Malmo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vesikari T, Ostergaard L, Beeslaar J, Absalon J, Eiden JJ, Jansen KU, Jones TR, Harris SL, Maansson R, Munson S, O'Neill RE, York LJ, Perez JL. Persistence and 4-year boosting of the bactericidal response elicited by two- and three-dose schedules of MenB-FHbp: A phase 3 extension study in adolescents. Vaccine. 2019 Mar 14;37(12):1710-1719. doi: 10.1016/j.vaccine.2018.11.073. Epub 2019 Feb 12. PMID 30770221
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1971033&StudyName=Duration%20of%20Immunity%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 698 participants enrolled in this extension study, who were enrolled in any 1 of the primary studies B1971010 (NCT01323270), B1971012 (NCT01299480), and B1971015 (NCT01461980).
Pre-assignment Details: This study consisted of 2 stages: Stage 1 and Booster stage. Only participants from primary studies B1971010 and B1971012 who received bivalent rLP2086 in the primary study and completed Stage 1 in this study, were eligible to participate in the booster stage.
Groups:
- Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule): Participants received quadrivalent meningococcal polysaccharide conjugate (MCV4) tetanus + acellular pertussis (Tdap) +Saline at Month 0, Saline only at Month 2 and 6 schedule in primary study B1971015 and were followed up for 48 months during the stage 1 of this study.
- Group 2: rLP2086 (0-, 1-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 1-, and 6-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study, and received intramuscular injection of 120 micrograms (mcg) of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Group 3: rLP2086 (0-, 2-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971010, B1971012 and B1971015 were included in this group, and were followed up for 48 months during the stage 1 of this study. Only participants from B1971010 and B1971012 studies received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Group 4: rLP2086 (0-and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0- and 6-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study, and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Group 5: rLP2086 (0- and 2-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0- and 2-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study, and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Group 6: rLP2086 (0- and 4-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0- and 4-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study, and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
Period: Stage 1 (48 Months)
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Started | 70 | 103 | 277 | 116 | 86 | 46
Safety Population (Participants who had at least 1 blood draw in this study.) | 70 | 101 | 277 | 116 | 86 | 46
Completed | 56 | 93 | 237 | 108 | 83 | 46
Not Completed | 14 | 10 | 40 | 8 | 3 | 0
Not completed — Lost to Follow-up | 3 | 4 | 12 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 1 | 0 | 1 | 2 | 0 | 0
Not completed — No longer willing to participate | 5 | 3 | 18 | 6 | 3 | 0
Not completed — Other than specified | 5 | 0 | 9 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0
Period: Booster Stage (26 Months)
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Started | 0 (Group1 participants (primary study B1971015)were not invited to participate in Booster stage (BS).) | 60 (BS was optional for eligible participants. Not all participants completing stage 1 continued to BS.) | 92 (BS was optional for eligible participants. Not all participants completing stage 1 continued to BS.) | 64 (BS was optional for eligible participants. Not all participants completing stage 1 continued to BS.) | 56 (BS was optional for eligible participants. Not all participants completing stage 1 continued to BS.) | 32 (BS was optional for eligible participants. Not all participants completing stage 1 continued to BS.)
Vaccinated | 0 | 59 | 92 | 64 | 54 | 32
Completed | 0 | 59 | 91 | 64 | 54 | 32
Not Completed | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Withdrawal before booster vaccination | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants enrolled in this study from primary studies B1971010, B1971012, and B1971015.
Groups:
- Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule): Participants received MCV4+Tdap+Saline at Month 0, Saline only at Month 2 and 6 schedule in primary study B1971015 and were followed up for 48 months during the stage 1 of this study.
- Total: Total of all reporting groups
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule) | Total
Number analyzed (Participants) | 70 | 103 | 277 | 116 | 86 | 46 | 698
Age, Continuous [Mean (Standard Deviation); unit: years] — The age of participants enrolled in B1971033 is the age of participants at Stage 1 enrollment.
  years | 11.7 (0.7) | 15.9 (2.2) | 14.3 (2.8) | 15.8 (2.1) | 16.1 (2.4) | 15.9 (2.1) | 14.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 55 | 144 | 67 | 38 | 26 | 362
  Male | 38 | 48 | 133 | 49 | 48 | 20 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 0 | 25 | 1 | 2 | 0 | 44
  Not Hispanic or Latino | 54 | 103 | 252 | 115 | 84 | 46 | 654
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59 | 103 | 256 | 115 | 85 | 46 | 664
  Black | 9 | 0 | 12 | 1 | 0 | 0 | 22
  Other | 2 | 0 | 8 | 0 | 1 | 0 | 11
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Stage 1 Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains at Month 6 (Visit 1) After Primary Vaccinations
Description: For immunogenicity assessment, serum bactericidal assay using human complement (hSBA) was performed with 4 primary Neisseria meningitidis serogroup B (MnB) test strains. Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 percent (%) confidence interval (CIs). LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44). Participants who received bivalent rLP2086 in primary study B1971012, entered in this study at Month 12 (Visit 2). Hence, no participants enrolled from primary study B1971012 had serology results at Month 6.
Time Frame: Month 6 (Visit 1 of study B1971033)
Population: Modified intent-to-treat (mITT) population included participants who had at least 1 valid and determinate assay result in Stage 1 of Study B1971033. Here, 'Number analyzed' signifies number of participants with valid and determinate hSBA titers for the given strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971010, received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately Month 48) in booster stage of study B1971033.
- Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule)): Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971015.
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule))
Number analyzed (Participants) | 70 | 40 | 123
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 7 | 37 | 18
  PMB80 (A22) | 14.3 [0.4 to 57.9] | 86.5 [71.2 to 95.5] | 83.3 [58.6 to 96.4]
  PMB2001 (A56): number analyzed (Participants) | 6 | 36 | 18
  PMB2001 (A56) | 16.7 [0.4 to 64.1] | 72.2 [54.8 to 85.8] | 88.9 [65.3 to 98.6]
  PMB2948 (B24): number analyzed (Participants) | 7 | 38 | 17
  PMB2948 (B24) | 0.0 [0.0 to 41.0] | 36.8 [21.8 to 54.0] | 35.3 [14.2 to 61.7]
  PMB2707 (B44): number analyzed (Participants) | 7 | 37 | 16
  PMB2707 (B44) | 0.0 [0.0 to 41.0] | 64.9 [47.5 to 79.8] | 56.3 [29.9 to 80.2]

2. Primary Outcome: Percentage of Participants in Stage 1 Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains at Month 12 (Visit 2) After Primary Vaccinations
Description: For immunogenicity assessment, hSBA was performed with 4 primary MnB test strains. Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 % CIs. LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: Month 12 (Visit 2 of study B1971033)
Population: mITT population included participants who had at least 1 valid and determinate assay result in Stage 1 of Study B1971033. Here, 'Number analyzed' signifies number of participants with valid and determinate hSBA titers for the given strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971012, received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately Month 48) in booster stage of study B1971033.
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule)) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 70 | 101 | 40 | 114 | 123 | 116 | 86 | 46
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 69 | 99 | 39 | 111 | 122 | 113 | 84 | 46
  PMB80 (A22) | 29.0 [18.7 to 41.2] | 41.4 [31.6 to 51.8] | 69.2 [52.4 to 83.0] | 45.0 [35.6 to 54.8] | 61.5 [52.2 to 70.1] | 36.3 [27.4 to 45.9] | 44.0 [33.2 to 55.3] | 41.3 [27.0 to 56.8]
  PMB2001 (A56): number analyzed (Participants) | 69 | 98 | 39 | 109 | 111 | 106 | 84 | 42
  PMB2001 (A56) | 17.4 [9.3 to 28.4] | 73.5 [63.6 to 81.9] | 66.7 [49.8 to 80.9] | 76.1 [67.0 to 83.8] | 63.1 [53.4 to 72.0] | 60.4 [50.4 to 69.7] | 69.0 [58.0 to 78.7] | 71.4 [55.4 to 84.3]
  PMB2948 (B24): number analyzed (Participants) | 70 | 98 | 40 | 108 | 121 | 103 | 82 | 46
  PMB2948 (B24) | 1.4 [0.0 to 7.7] | 40.8 [31.0 to 51.2] | 37.5 [22.7 to 54.2] | 49.1 [39.3 to 58.9] | 24.0 [16.7 to 32.6] | 36.9 [27.6 to 47.0] | 41.5 [30.7 to 52.9] | 37.0 [23.2 to 52.5]
  PMB2707 (B44): number analyzed (Participants) | 70 | 100 | 40 | 111 | 120 | 115 | 85 | 45
  PMB2707 (B44) | 1.4 [0.0 to 7.7] | 24.0 [16.0 to 33.6] | 47.5 [31.5 to 63.9] | 22.5 [15.1 to 31.4] | 32.5 [24.2 to 41.7] | 16.5 [10.3 to 24.6] | 21.2 [13.1 to 31.4] | 22.2 [11.2 to 37.1]

3. Primary Outcome: Percentage of Participants in Stage 1 Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains at Month 18 (Visit 3) After Primary Vaccinations
Description: as for outcome 2
Time Frame: Month 18 (Visit 3 of study B1971033)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule)) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 70 | 101 | 40 | 114 | 123 | 116 | 86 | 46
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 69 | 97 | 38 | 112 | 117 | 111 | 85 | 45
  PMB80 (A22) | 23.2 [13.9 to 34.9] | 37.1 [27.5 to 47.5] | 57.9 [40.8 to 73.7] | 44.6 [35.2 to 54.3] | 51.3 [41.9 to 60.6] | 47.7 [38.2 to 57.4] | 47.1 [36.1 to 58.2] | 51.1 [35.8 to 66.3]
  PMB2001 (A56): number analyzed (Participants) | 67 | 94 | 39 | 106 | 114 | 102 | 83 | 43
  PMB2001 (A56) | 11.9 [5.3 to 22.2] | 64.9 [54.4 to 74.5] | 56.4 [39.6 to 72.2] | 72.6 [63.1 to 80.9] | 53.5 [43.9 to 62.9] | 57.8 [47.7 to 67.6] | 62.7 [51.3 to 73.0] | 62.8 [46.7 to 77.0]
  PMB2948 (B24): number analyzed (Participants) | 69 | 96 | 38 | 109 | 113 | 105 | 81 | 44
  PMB2948 (B24) | 5.8 [1.6 to 14.2] | 45.8 [35.6 to 56.3] | 39.5 [24.0 to 56.6] | 46.8 [37.2 to 56.6] | 23.9 [16.4 to 32.8] | 31.4 [22.7 to 41.2] | 39.5 [28.8 to 51.0] | 50.0 [34.6 to 65.4]
  PMB2707 (B44): number analyzed (Participants) | 69 | 98 | 38 | 110 | 115 | 113 | 86 | 46
  PMB2707 (B44) | 0.0 [0.0 to 5.2] | 26.5 [18.1 to 36.4] | 31.6 [17.5 to 48.7] | 18.2 [11.5 to 26.7] | 29.6 [21.4 to 38.8] | 15.9 [9.7 to 24.0] | 24.4 [15.8 to 34.9] | 28.3 [16.0 to 43.5]

4. Primary Outcome: Percentage of Participants in Stage 1 Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains at Month 24 (Visit 4) After Primary Vaccinations
Description: as for outcome 2
Time Frame: Month 24 (Visit 4 of study B1971033)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule)) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 70 | 101 | 40 | 114 | 123 | 116 | 86 | 46
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 68 | 98 | 38 | 107 | 115 | 109 | 84 | 46
  PMB80 (A22) | 17.6 [9.5 to 28.8] | 34.7 [25.4 to 45.0] | 50.0 [33.4 to 66.6] | 40.2 [30.8 to 50.1] | 49.6 [40.1 to 59.0] | 42.2 [32.8 to 52.0] | 44.0 [33.2 to 55.3] | 39.1 [25.1 to 54.6]
  PMB2001 (A56): number analyzed (Participants) | 66 | 91 | 38 | 102 | 110 | 104 | 80 | 45
  PMB2001 (A56) | 3.0 [0.4 to 10.5] | 69.2 [58.7 to 78.5] | 57.9 [40.8 to 73.7] | 68.6 [58.7 to 77.5] | 36.4 [27.4 to 46.1] | 53.8 [43.8 to 63.7] | 58.8 [47.2 to 69.6] | 60.0 [44.3 to 74.3]
  PMB2948 (B24): number analyzed (Participants) | 68 | 93 | 38 | 107 | 112 | 110 | 83 | 45
  PMB2948 (B24) | 4.4 [0.9 to 12.4] | 43.0 [32.8 to 53.7] | 39.5 [24.0 to 56.6] | 43.0 [33.5 to 52.9] | 25.9 [18.1 to 35.0] | 31.8 [23.3 to 41.4] | 37.3 [27.0 to 48.7] | 51.1 [35.8 to 66.3]
  PMB2707 (B44): number analyzed (Participants) | 67 | 97 | 39 | 109 | 114 | 108 | 83 | 46
  PMB2707 (B44) | 3.0 [0.4 to 10.4] | 23.7 [15.7 to 33.4] | 38.5 [23.4 to 55.4] | 18.3 [11.6 to 26.9] | 27.2 [19.3 to 36.3] | 15.7 [9.4 to 24.0] | 22.9 [14.4 to 33.4] | 28.3 [16.0 to 43.5]

5. Primary Outcome: Percentage of Participants in Stage 1 Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains at Month 36 (Visit 5) After Primary Vaccinations
Description: as for outcome 2
Time Frame: Month 36 (Visit 5 of study B1971033)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule)) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 70 | 101 | 40 | 114 | 123 | 116 | 86 | 46
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 58 | 96 | 38 | 102 | 107 | 108 | 82 | 44
  PMB80 (A22) | 27.6 [16.7 to 40.9] | 41.7 [31.7 to 52.2] | 60.5 [43.4 to 76.0] | 39.2 [29.7 to 49.4] | 49.5 [39.7 to 59.4] | 42.6 [33.1 to 52.5] | 42.7 [31.8 to 54.1] | 34.1 [20.5 to 49.9]
  PMB2001 (A56): number analyzed (Participants) | 57 | 94 | 37 | 92 | 103 | 99 | 81 | 42
  PMB2001 (A56) | 7.0 [1.9 to 17.0] | 58.5 [47.9 to 68.6] | 54.1 [36.9 to 70.5] | 67.4 [56.8 to 76.8] | 35.0 [25.8 to 45.0] | 58.6 [48.2 to 68.4] | 59.3 [47.8 to 70.1] | 50.0 [34.2 to 65.8]
  PMB2948 (B24): number analyzed (Participants) | 59 | 93 | 36 | 100 | 103 | 107 | 81 | 43
  PMB2948 (B24) | 3.4 [0.4 to 11.7] | 41.9 [31.8 to 52.6] | 38.9 [23.1 to 56.5] | 42.0 [32.2 to 52.3] | 30.1 [21.5 to 39.9] | 33.6 [24.8 to 43.4] | 48.1 [36.9 to 59.5] | 41.9 [27.0 to 57.9]
  PMB2707 (B44): number analyzed (Participants) | 59 | 97 | 39 | 103 | 103 | 109 | 83 | 44
  PMB2707 (B44) | 1.7 [0.0 to 9.1] | 21.6 [13.9 to 31.2] | 33.3 [19.1 to 50.2] | 16.5 [9.9 to 25.1] | 24.3 [16.4 to 33.7] | 20.2 [13.1 to 28.9] | 21.7 [13.4 to 32.1] | 18.2 [8.2 to 32.7]

6. Primary Outcome: Percentage of Participants in Stage 1 Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains at Month 48 (Visit 6) After Primary Vaccinations
Description: as for outcome 2
Time Frame: Month 48 (Visit 6 of study B1971033)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971015 received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately Month 48) in booster stage of this study.
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3c: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 70 | 101 | 40 | 114 | 123 | 116 | 86 | 46
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 55 | 90 | 35 | 100 | 101 | 101 | 81 | 46
  PMB80 (A22) | 16.4 [7.8 to 28.8] | 41.1 [30.8 to 52.0] | 51.4 [34.0 to 68.6] | 43.0 [33.1 to 53.3] | 34.7 [25.5 to 44.8] | 39.6 [30.0 to 49.8] | 45.7 [34.6 to 57.1] | 41.3 [27.0 to 56.8]
  PMB2001 (A56): number analyzed (Participants) | 51 | 85 | 33 | 99 | 94 | 99 | 75 | 46
  PMB2001 (A56) | 2.0 [0.0 to 10.4] | 47.1 [36.1 to 58.2] | 42.4 [25.5 to 60.8] | 58.6 [48.2 to 68.4] | 30.9 [21.7 to 41.2] | 57.6 [47.2 to 67.5] | 61.3 [49.4 to 72.4] | 47.8 [32.9 to 63.1]
  PMB2948 (B24): number analyzed (Participants) | 56 | 90 | 34 | 98 | 101 | 105 | 82 | 45
  PMB2948 (B24) | 7.1 [2.0 to 17.3] | 41.1 [30.8 to 52.0] | 50.0 [32.4 to 67.6] | 40.8 [31.0 to 51.2] | 23.8 [15.9 to 33.3] | 30.5 [21.9 to 40.2] | 45.1 [34.1 to 56.5] | 42.2 [27.7 to 57.8]
  PMB2707 (B44): number analyzed (Participants) | 56 | 92 | 34 | 100 | 100 | 106 | 82 | 46
  PMB2707 (B44) | 3.6 [0.4 to 12.3] | 20.7 [12.9 to 30.4] | 41.2 [24.6 to 59.3] | 18.0 [11.0 to 26.9] | 23.0 [15.2 to 32.5] | 18.9 [11.9 to 27.6] | 24.4 [15.6 to 35.1] | 23.9 [12.6 to 38.8]

7. Primary Outcome: Percentage of Booster Stage Participants Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains 1 Month After Last Vaccination in Primary Study
Description: For immunogenicity assessment, hSBA was performed with 4 primary MnB test strains. Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 % CIs. LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44). Participants of Group 3c (participants from primary study B1971015) were not continued in booster stage.
Time Frame: 1 month after last vaccination in primary study
Population: Evaluable population:eligible participants who received scheduled investigational products, received no prohibited vaccines or treatment, had pre and post vaccination blood drawn with valid,determinate assay results and had no important protocol deviation. 'Number analyzed'=number of participants with valid,determinate hSBA titers for given strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 31 | 58 | 62 | 54 | 32
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 59 | 31 | 57 | 61 | 54 | 32
  PMB80 (A22) | 89.8 [79.2 to 96.2] | 100.0 [88.8 to 100.0] | 91.2 [80.7 to 97.1] | 98.4 [91.2 to 100.0] | 77.8 [64.4 to 88.0] | 84.4 [67.2 to 94.7]
  PMB2001 (A56): number analyzed (Participants) | 58 | 31 | 57 | 62 | 54 | 32
  PMB2001 (A56) | 100.0 [93.8 to 100.0] | 100.0 [88.8 to 100.0] | 98.2 [90.6 to 100.0] | 98.4 [91.3 to 100.0] | 100.0 [93.4 to 100.0] | 96.9 [83.8 to 99.9]
  PMB2948 (B24): number analyzed (Participants) | 59 | 31 | 58 | 60 | 52 | 29
  PMB2948 (B24) | 88.1 [77.1 to 95.1] | 93.5 [78.6 to 99.2] | 91.4 [81.0 to 97.1] | 85.0 [73.4 to 92.9] | 71.2 [56.9 to 82.9] | 79.3 [60.3 to 92.0]
  PMB2707 (B44): number analyzed (Participants) | 58 | 31 | 57 | 60 | 52 | 32
  PMB2707 (B44) | 86.2 [74.6 to 93.9] | 96.8 [83.3 to 99.9] | 89.5 [78.5 to 96.0] | 81.7 [69.6 to 90.5] | 73.1 [59.0 to 84.4] | 87.5 [71.0 to 96.5]

8. Primary Outcome: Percentage of Booster Stage Participants Achieving hSBA Titer Level (>=) Lower Limit of Quantitation for Each of the 4 Primary Strains Before Booster Vaccination (48 Months After Last Vaccination in Primary Study [Visit 6])
Description: as for outcome 7
Time Frame: Visit 6 of study B1971033 (48 months after last vaccination in primary study)
Population: Evaluable population:eligible participants who received scheduled investigational products, received no prohibited vaccines or treatment, had pre and post vaccination blood drawn with valid, determinate assay results and had no important protocol deviation. 'Number analyzed'=number of participants with valid,determinatehSBA titers for given strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 31 | 58 | 62 | 54 | 32
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 59 | 31 | 57 | 61 | 54 | 31
  PMB80 (A22) | 49.2 [35.9 to 62.5] | 48.4 [30.2 to 66.9] | 56.1 [42.4 to 69.3] | 55.7 [42.4 to 68.5] | 57.4 [43.2 to 70.8] | 48.4 [30.2 to 66.9]
  PMB2001 (A56): number analyzed (Participants) | 53 | 29 | 55 | 62 | 52 | 30
  PMB2001 (A56) | 43.4 [29.8 to 57.7] | 41.4 [23.5 to 61.1] | 56.4 [42.3 to 69.7] | 43.5 [31.0 to 56.7] | 51.9 [37.6 to 66.0] | 43.3 [25.5 to 62.6]
  PMB2948 (B24): number analyzed (Participants) | 59 | 30 | 57 | 62 | 54 | 31
  PMB2948 (B24) | 40.7 [28.1 to 54.3] | 46.7 [28.3 to 65.7] | 49.1 [35.6 to 62.7] | 40.3 [28.1 to 53.6] | 46.3 [32.6 to 60.4] | 45.2 [27.3 to 64.0]
  PMB2707 (B44): number analyzed (Participants) | 57 | 30 | 57 | 62 | 53 | 32
  PMB2707 (B44) | 36.8 [24.4 to 50.7] | 33.3 [17.3 to 52.8] | 35.1 [22.9 to 48.9] | 12.9 [5.7 to 23.9] | 37.7 [24.8 to 52.1] | 34.4 [18.6 to 53.2]

9. Primary Outcome: Percentage of Participants Achieving hSBA Titer Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains 1 Month After the Booster Vaccination (Visit 8)
Description: as for outcome 7
Time Frame: Visit 8 (1 month following the booster vaccination on Month 49)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 31 | 58 | 62 | 54 | 32
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 59 | 31 | 58 | 60 | 53 | 32
  PMB80 (A22) | 100.0 [93.9 to 100.0] | 96.8 [83.3 to 99.9] | 100.0 [93.8 to 100.0] | 96.7 [88.5 to 99.6] | 98.1 [89.9 to 100.0] | 100.0 [89.1 to 100.0]
  PMB2001 (A56): number analyzed (Participants) | 57 | 30 | 56 | 62 | 51 | 32
  PMB2001 (A56) | 100.0 [93.7 to 100.0] | 100.0 [88.4 to 100.0] | 100.0 [93.6 to 100.0] | 98.4 [91.3 to 100.0] | 100.0 [93.0 to 100.0] | 100.0 [89.1 to 100.0]
  PMB2948 (B24): number analyzed (Participants) | 58 | 31 | 57 | 62 | 54 | 32
  PMB2948 (B24) | 100.0 [93.8 to 100.0] | 96.8 [83.3 to 99.9] | 100.0 [93.7 to 100.0] | 96.8 [88.8 to 99.6] | 94.4 [84.6 to 98.8] | 100.0 [89.1 to 100.0]
  PMB2707 (B44): number analyzed (Participants) | 59 | 31 | 58 | 61 | 53 | 32
  PMB2707 (B44) | 100.0 [93.9 to 100.0] | 100.0 [88.8 to 100.0] | 100.0 [93.8 to 100.0] | 93.4 [84.1 to 98.2] | 100.0 [93.3 to 100.0] | 100.0 [89.1 to 100.0]

10. Primary Outcome: Percentage of Participants Achieving hSBATiter Level Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains 12 Months After the Booster Vaccination(Visit 10)
Description: as for outcome 7
Time Frame: Visit 10 (12 months following the booster vaccination on Month 60)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3a: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 31 | 58 | 62 | 54 | 32
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 58 | 28 | 54 | 60 | 51 | 31
  PMB80 (A22) | 74.1 [61.0 to 84.7] | 89.3 [71.8 to 97.7] | 77.8 [64.4 to 88.0] | 80.0 [67.7 to 89.2] | 82.4 [69.1 to 91.6] | 96.8 [83.3 to 99.9]
  PMB2001 (A56): number analyzed (Participants) | 55 | 24 | 55 | 59 | 50 | 32
  PMB2001 (A56) | 90.9 [80.0 to 97.0] | 87.5 [67.6 to 97.3] | 89.1 [77.8 to 95.9] | 81.4 [69.1 to 90.3] | 74.0 [59.7 to 85.4] | 100.0 [89.1 to 100.0]
  PMB2948 (B24): number analyzed (Participants) | 58 | 30 | 54 | 62 | 49 | 32
  PMB2948 (B24) | 65.5 [51.9 to 77.5] | 66.7 [47.2 to 82.7] | 74.1 [60.3 to 85.0] | 77.4 [65.0 to 87.1] | 65.3 [50.4 to 78.3] | 84.4 [67.2 to 94.7]
  PMB2707 (B44): number analyzed (Participants) | 56 | 30 | 53 | 61 | 52 | 30
  PMB2707 (B44) | 75.0 [61.6 to 85.6] | 76.7 [57.7 to 90.1] | 81.1 [68.0 to 90.6] | 59.0 [45.7 to 71.4] | 78.8 [65.3 to 88.9] | 93.3 [77.9 to 99.2]

11. Primary Outcome: Percentage of Participants Achieving hSBA Titer Level Greater Than or Equal to(>=) Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Strains 26 Months After the Booster Vaccination(Visit 11)
Description: For immunogenicity assessment, hSBA was performed with 4 primary MnB test strains. Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 % CIs. LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44). Participants of Group 3c (participants from primary study B1971015) were not continued in booster stage. only participants who received bivalent rLP2086 in primary study B1971010 were not analysed for this endpoint. Only participants who received bivalent rLP2086 in primary study B1971012 on a 0-, 2-, and 6-month or a 0- and 6-month vaccination schedule were eligible to be followed for 26 months after booster vaccination
Time Frame: Visit 11 (26 months following the booster vaccination on Month 74)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule)
Number analyzed (Participants) | 58 | 62
percentage of participants
  PMB80 (A22): number analyzed (Participants) | 34 | 42
  PMB80 (A22) | 73.5 [55.6 to 87.1] | 61.9 [45.6 to 76.4]
  PMB2001 (A56): number analyzed (Participants) | 29 | 40
  PMB2001 (A56) | 82.8 [64.2 to 94.2] | 57.5 [40.9 to 73.0]
  PMB2948 (B24): number analyzed (Participants) | 33 | 42
  PMB2948 (B24) | 78.8 [61.1 to 91.0] | 59.5 [43.3 to 74.4]
  PMB2707 (B44): number analyzed (Participants) | 33 | 43
  PMB2707 (B44) | 66.7 [48.2 to 82.0] | 62.8 [46.7 to 77.0]

12. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Booster Vaccination
Description: Local reactions were collected by using an e-diary and included pain at injection site, redness and swelling. Redness and swelling were graded as: none (0-2.0 centimetre [cm]), mild (2.5-5.0 cm), moderate (greater than [>] 5.0-10.0 cm) and severe (>10.0 cm). Pain was graded as: mild (does not interfere with activity), moderate (Interferes with activity) and severe (prevents daily activity).
Time Frame: Within 7 days after booster vaccination on Month 48
Population: Booster stage safety population included all participants who had received the booster vaccination (Bivalent rLP2086) and for whom safety data was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants
  Pain at injection site:Any | 91.5 [81.3 to 97.2] | 93.5 [86.3 to 97.6] | 89.1 [78.8 to 95.5] | 88.9 [77.4 to 95.8] | 84.4 [67.2 to 94.7]
  Pain at injection site:Mild | 37.3 [25.0 to 50.9] | 29.3 [20.3 to 39.8] | 28.1 [17.6 to 40.8] | 35.2 [22.7 to 49.4] | 25.0 [11.5 to 43.4]
  Pain at injection site:Moderate | 40.7 [28.1 to 54.3] | 54.3 [43.6 to 64.8] | 51.6 [38.7 to 64.2] | 44.4 [30.9 to 58.6] | 46.9 [29.1 to 65.3]
  Pain at injection site:Severe | 13.6 [6.0 to 25.0] | 9.8 [4.6 to 17.8] | 9.4 [3.5 to 19.3] | 9.3 [3.1 to 20.3] | 12.5 [3.5 to 29.0]
  Redness:Any | 20.3 [11.0 to 32.8] | 20.7 [12.9 to 30.4] | 20.3 [11.3 to 32.2] | 27.8 [16.5 to 41.6] | 6.3 [0.8 to 20.8]
  Redness:Mild | 6.8 [1.9 to 16.5] | 5.4 [1.8 to 12.2] | 10.9 [4.5 to 21.2] | 5.6 [1.2 to 15.4] | 3.1 [0.1 to 16.2]
  Redness:Moderate | 11.9 [4.9 to 22.9] | 10.9 [5.3 to 19.1] | 7.8 [2.6 to 17.3] | 16.7 [7.9 to 29.3] | 3.1 [0.1 to 16.2]
  Redness:Severe | 1.7 [0.0 to 9.1] | 4.3 [1.2 to 10.8] | 1.6 [0.0 to 8.4] | 5.6 [1.2 to 15.4] | 0.0 [0.0 to 10.9]
  Swelling:Any | 18.6 [9.7 to 30.9] | 20.7 [12.9 to 30.4] | 17.2 [8.9 to 28.7] | 14.8 [6.6 to 27.1] | 9.4 [2.0 to 25.0]
  Swelling:Mild | 11.9 [4.9 to 22.9] | 8.7 [3.8 to 16.4] | 10.9 [4.5 to 21.2] | 3.7 [0.5 to 12.7] | 9.4 [2.0 to 25.0]
  Swelling:Moderate | 6.8 [1.9 to 16.5] | 10.9 [5.3 to 19.1] | 6.3 [1.7 to 15.2] | 11.1 [4.2 to 22.6] | 0.0 [0.0 to 10.9]
  Swelling:Severe | 0.0 [0.0 to 6.1] | 1.1 [0.0 to 5.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]

13. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Booster Vaccination
Description: Systemic reactions included: fever, vomiting, diarrhea, headache, fatigue, chills, muscle pain other than muscle pain at the injection site and joint pain, all other systemic reactions were recorded by using an e-diary. Fever was categorized as: 38.0 to 38.4 degree Celsius (C), 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and > 40.0 degree C. Vomiting was graded as: mild (1 to 2 times in 24 hours [hrs]), moderate (>2 times in 24 hrs) and severe (requires intravenous [IV] hydration); Diarrhea was graded as: mild (2 to 3 loose stools in 24 hrs), moderate (4 to 5 loose stools in 24 hrs) and severe (6 or more loose stools in 24 hrs); Headache, fatigue, chills, muscle pain and joint pain was graded as: mild (does not interfere with daily activities), moderate (some interference with activity) and severe (prevents daily routine activity).
Time Frame: Within 7 days after booster vaccination on Month 48
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants
  Fever >=38 degrees C | 5.1 [1.1 to 14.1] | 1.1 [0.0 to 5.9] | 4.7 [1.0 to 13.1] | 1.9 [0.0 to 9.9] | 3.1 [0.1 to 16.2]
  Fever 38.0 to <38.5 degrees C | 5.1 [1.1 to 14.1] | 1.1 [0.0 to 5.9] | 3.1 [0.4 to 10.8] | 0.0 [0.0 to 6.6] | 3.1 [0.1 to 16.2]
  Fever 38.5 to <39.0 degrees C | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 1.6 [0.0 to 8.4] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  Fever 39.0 to 40.0 degrees C | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Fever >40.0 degrees C | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Vomiting:Any | 1.7 [0.0 to 9.1] | 3.3 [0.7 to 9.2] | 3.1 [0.4 to 10.8] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  Vomiting:Mild | 1.7 [0.0 to 9.1] | 3.3 [0.7 to 9.2] | 1.6 [0.0 to 8.4] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  Vomiting:Moderate | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 1.6 [0.0 to 8.4] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Vomiting:Severe | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Diarrhea:Any | 10.2 [3.8 to 20.8] | 13.0 [6.9 to 21.7] | 4.7 [1.0 to 13.1] | 5.6 [1.2 to 15.4] | 18.8 [7.2 to 36.4]
  Diarrhea:Mild | 8.5 [2.8 to 18.7] | 12.0 [6.1 to 20.4] | 3.1 [0.4 to 10.8] | 5.6 [1.2 to 15.4] | 18.8 [7.2 to 36.4]
  Diarrhea:Moderate | 1.7 [0.0 to 9.1] | 1.1 [0.0 to 5.9] | 1.6 [0.0 to 8.4] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Diarrhea:Severe | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Headache:Any | 50.8 [37.5 to 64.1] | 47.8 [37.3 to 58.5] | 56.3 [43.3 to 68.6] | 48.1 [34.3 to 62.2] | 37.5 [21.1 to 56.3]
  Headache:Mild | 30.5 [19.2 to 43.9] | 28.3 [19.4 to 38.6] | 35.9 [24.3 to 48.9] | 22.2 [12.0 to 35.6] | 25.0 [11.5 to 43.4]
  Headache:Moderate | 20.3 [11.0 to 32.8] | 18.5 [11.1 to 27.9] | 20.3 [11.3 to 32.2] | 25.9 [15.0 to 39.7] | 12.5 [3.5 to 29.0]
  Headache:Severe | 0.0 [0.0 to 6.1] | 1.1 [0.0 to 5.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  Fatigue:Any | 62.7 [49.1 to 75.0] | 60.9 [50.1 to 70.9] | 62.5 [49.5 to 74.3] | 51.9 [37.8 to 65.7] | 65.6 [46.8 to 81.4]
  Fatigue:Mild | 27.1 [16.4 to 40.3] | 27.2 [18.4 to 37.4] | 35.9 [24.3 to 48.9] | 24.1 [13.5 to 37.6] | 31.3 [16.1 to 50.0]
  Fatigue:Moderate | 32.2 [20.6 to 45.6] | 31.5 [22.2 to 42.0] | 23.4 [13.8 to 35.7] | 24.1 [13.5 to 37.6] | 31.3 [16.1 to 50.0]
  Fatigue:Severe | 3.4 [0.4 to 11.7] | 2.2 [0.3 to 7.6] | 3.1 [0.4 to 10.8] | 3.7 [0.5 to 12.7] | 3.1 [0.1 to 16.2]
  Chills:Any | 23.7 [13.6 to 36.6] | 31.5 [22.2 to 42.0] | 20.3 [11.3 to 32.2] | 18.5 [9.3 to 31.4] | 28.1 [13.7 to 46.7]
  Chills:Mild | 13.6 [6.0 to 25.0] | 20.7 [12.9 to 30.4] | 12.5 [5.6 to 23.2] | 9.3 [3.1 to 20.3] | 18.8 [7.2 to 36.4]
  Chills:Moderate | 10.2 [3.8 to 20.8] | 9.8 [4.6 to 17.8] | 7.8 [2.6 to 17.3] | 7.4 [2.1 to 17.9] | 9.4 [2.0 to 25.0]
  Chills:Severe | 0.0 [0.0 to 6.1] | 1.1 [0.0 to 5.9] | 0.0 [0.0 to 5.6] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  Muscle pain:Any | 22.0 [12.3 to 34.7] | 29.3 [20.3 to 39.8] | 18.8 [10.1 to 30.5] | 24.1 [13.5 to 37.6] | 15.6 [5.3 to 32.8]
  Muscle pain: Mild | 16.9 [8.4 to 29.0] | 15.2 [8.6 to 24.2] | 7.8 [2.6 to 17.3] | 14.8 [6.6 to 27.1] | 6.3 [0.8 to 20.8]
  Muscle pain:Moderate | 5.1 [1.1 to 14.1] | 13.0 [6.9 to 21.7] | 7.8 [2.6 to 17.3] | 5.6 [1.2 to 15.4] | 9.4 [2.0 to 25.0]
  Muscle pain:Severe | 0.0 [0.0 to 6.1] | 1.1 [0.0 to 5.9] | 3.1 [0.4 to 10.8] | 3.7 [0.5 to 12.7] | 0.0 [0.0 to 10.9]
  Joint pain:Any | 11.9 [4.9 to 22.9] | 16.3 [9.4 to 25.5] | 14.1 [6.6 to 25.0] | 18.5 [9.3 to 31.4] | 21.9 [9.3 to 40.0]
  Joint pain:Mild | 8.5 [2.8 to 18.7] | 9.8 [4.6 to 17.8] | 7.8 [2.6 to 17.3] | 7.4 [2.1 to 17.9] | 12.5 [3.5 to 29.0]
  Joint pain:Moderate | 3.4 [0.4 to 11.7] | 6.5 [2.4 to 13.7] | 4.7 [1.0 to 13.1] | 9.3 [3.1 to 20.3] | 9.4 [2.0 to 25.0]
  Joint pain:Severe | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 1.6 [0.0 to 8.4] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  Use of antipyretic medication | 10.2 [3.8 to 20.8] | 14.1 [7.7 to 23.0] | 7.8 [2.6 to 17.3] | 13.0 [5.4 to 24.9] | 6.3 [0.8 to 20.8]

14. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE), Serious Adverse Event (SAE), Newly Diagnosed Chronic Medical Condition (NDCMC) and Medically Attended Adverse Event (MAE) From Booster Vaccination Phase (Visit 7 to Visit 8)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both non-serious AEs and serious adverse events (SAEs). An NDCMC was defined as a disease or medical condition, that was not identified previously and that was expected to be persistent or otherwise long-lasting in its effects. The investigator determined if the AE was an NDCMC. An MAE was defined as a non serious AE (AE other than SAE) that resulted in an evaluation at a medical facility.
Time Frame: From Visit 7 (Month 48) to Visit 8 (Month 49) in Booster stage
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants
  AE | 6.8 [1.9 to 16.5] | 8.7 [3.8 to 16.4] | 12.5 [5.6 to 23.2] | 3.7 [0.5 to 12.7] | 12.5 [3.5 to 29.0]
  SAE | 0.0 [0.0 to 6.1] | 1.1 [0.0 to 5.9] | 0.0 [0.0 to 5.6] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  NDCMC | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  MAE | 5.1 [1.1 to 14.1] | 4.3 [1.2 to 10.8] | 4.7 [1.0 to 13.1] | 0.0 [0.0 to 6.6] | 3.1 [0.1 to 16.2]

15. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) and Medically Attended Adverse Event (MAE) From Booster Follow-Up Phase (Visit 8 to Visit 9)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An MAE was defined as a non serious AE (AE other than SAE) that resulted in an evaluation at a medical facility.
Time Frame: Visit 8 (Month 49) to Visit 9 (Month 54) in Booster stage
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants
  SAE | 1.7 [0.0 to 9.1] | 0.0 [0.0 to 3.9] | 3.1 [0.4 to 10.8] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]
  MAE | 28.8 [17.8 to 42.1] | 12.0 [6.1 to 20.4] | 10.9 [4.5 to 21.2] | 11.1 [4.2 to 22.6] | 21.9 [9.3 to 40.0]

16. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) and Medically Attended Adverse Event (MAE) From Booster Vaccination Through 6 Months After Booster Vaccination (Visit 7 to Visit 9)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An MAE was defined as a nonserious AE (AE other than SAE) that resulted in an evaluation at a medical facility.
Time Frame: From Visit 7 (time of booster vaccination, Month 48) to Visit 9 (6 months after booster vaccination, Month 54)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants
  SAE | 1.7 [0.0 to 9.1] | 1.1 [0.0 to 5.9] | 3.1 [0.4 to 10.8] | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 10.9]
  MAE | 32.2 [20.6 to 45.6] | 15.2 [8.6 to 24.2] | 15.6 [7.8 to 26.9] | 11.1 [4.2 to 22.6] | 25.0 [11.5 to 43.4]

17. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition;(NDCMC) From the 6-Month Safety Telephone Call in the Primary Study Through 48 Months After the Last Dose in the Primary Study (Visit 6 in Stage 1)
Description: An NDCMC was defined as a disease or medical condition, that was not identified previously and that was expected to be persistent or otherwise long-lasting in its effects. The investigator determined if the AE was an NDCMC.
Time Frame: Visit 1 of B1971033 (6-month safety telephone call after last dose in primary study) to Visit 6 of B1971033 (6 months after last primary dose to 48 months after last primary dose in primary study)
Population: Stage 1 safety population included all participants who had at least 1 blood draw in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1:MCV4+Tdap+Saline (0-, 2-, and 6-Month Schedule) | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 70 | 101 | 277 | 116 | 86 | 46
percentage of participants | 5.7 [1.6 to 14.0] | 5.0 [1.6 to 11.2] | 2.2 [0.8 to 4.7] | 2.6 [0.5 to 7.4] | 2.3 [0.3 to 8.1] | 2.2 [0.1 to 11.5]

18. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) From 1 Month After Booster Vaccination Through 12 Months After Booster Vaccination (Visit 8 to Visit 10)
Description: as for outcome 17
Time Frame: From Visit 8 (1 month after booster vaccination, Month 49) to Visit 10 (12 months after booster vaccination, Month 60)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants | 1.7 [0.0 to 9.1] | 2.2 [0.3 to 7.6] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]

19. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) From Booster Stage Vaccination Through 12 Months After Booster Vaccination (Visit 7 to Visit 10)
Description: as for outcome 17
Time Frame: From Visit 7 (time of booster vaccination, Month 48) to Visit 10 (12 months after booster vaccination, Month 60)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants | 1.7 [0.0 to 9.1] | 2.2 [0.3 to 7.6] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 10.9]

20. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition (NDCMC) From 1 Month After Booster Vaccination Through 26 Months After Booster Vaccination (Visit 8 to Visit 11)
Description: An NDCMC was defined as a disease or medical condition, that was not identified previously and that was expected to be persistent or otherwise long-lasting in its effects. The investigator determined if the AE was an NDCMC. Participants who received bivalent rLP2086 in primary study B1971012 on a 0-, 2-, and 6-month or a 0- and 6-month vaccination schedule were eligible to be follow up for 26 months after booster vaccination.
Time Frame: From Visit 8 (1 month after booster vaccination, Month 49) to Visit 11 (26 months after booster vaccination, Month 74)
Population: Booster stage safety population included all participants who had received the booster vaccination (bivalent rLP2086) and for whom safety data was available. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule)
Number analyzed (Participants) | 37 | 49
percentage of participants | 5.4 [0.7 to 18.2] | 0.0 [0.0 to 7.3]

21. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition (NDCMC) From Booster Vaccine Through 26 Months After Booster Vaccination (Visit 7 to Visit 11)
Description: as for outcome 20
Time Frame: From Visit 7 (time of booster vaccination, Month 48) to Visit 11 (26 months after booster vaccination, Month 74)
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3b: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule)
Number analyzed (Participants) | 37 | 49
percentage of participants | 5.4 [0.7 to 18.2] | 0.0 [0.0 to 7.3]

22. Primary Outcome: Percentage of Participants With at Least 1 Immediate Adverse Event (AE) After Booster Vaccination
Description: Immediate AE was defined as AEs occurring within the first 30 minutes after investigational product administration. An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Within 30 minutes after Booster Vaccination in Month 48
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 59 | 92 | 64 | 54 | 32
percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

23. Primary Outcome: Number of Days Participants Missed Work or School Due to AE From Booster Vaccination Through 6 Months After Booster Vaccination (Visit 7 Through Visit 9)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Number of days participants missed work or school due to AE occurred following booster vaccination were reported here.
Time Frame: From Visit 7 (time of booster vaccination, Month 48) Through Visit 9 (6 months after booster vaccination, Month 54)
Population: Booster stage safety population included all participants who had received the booster vaccination (bivalent rLP2086) and for whom safety data was available. Here, "Overall number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Group 4: rLP2086 (0-and 6-Month Schedule) | Group 5: rLP2086 (0- and 2-Month Schedule) | Group 6: rLP2086 (0- and 4-Month Schedule)
Number analyzed (Participants) | 12 | 8 | 8 | 3 | 6
days | 17.5 (28.14) | 12.4 (9.72) | 10.1 (9.14) | 3.0 (2.65) | 4.8 (2.56)

ADVERSE EVENTS:
Time Frame: SAEs and Non SAEs: Visit 7 (Booster vaccination, Month 48) to Visit 11 (Month 74) [26 months]. Local reactions and systemic events: Recorded by participants in e-diary from Day 1 to Day 7 after booster vaccination in Month 48.
Description: AEs were reported only for those participants who had received the booster vaccination (bivalent rLP2086) and for whom safety information was available for disclosure. SAEs were not collected for stage 1 of the study.
Groups:
- Stage1,Group 1:MCV4+Tdap+Saline (0-,2-,and 6-Month Schedule):: Participants received MCV4+Tdap+Saline at Month 0, Saline only at Month 2 and 6 schedule in primary study B1971015 and were followed up for 48 months during the stage 1 of this study.
- Stage 1, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule):: Participants who received bivalent rLP2086 vaccine on 0-, 1-, and 6-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study.
- Stage 1, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule):: Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971010, B1971012 and B1971015 were included in this group, and were followed up for 48 months during the stage 1 of this study.
- Stage 1, Group 4: rLP2086 (0-and 6-Month Schedule):: Participants who received bivalent rLP2086 vaccine on 0- and 6-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study.
- Stage 1, Group 5: rLP2086 (0- and 2-Month Schedule):: Participants who received bivalent rLP2086 vaccine on 0- and 2-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study.
- Stage 1,Group 6: rLP2086 (0- and 4-Month Schedule):: Participants who received bivalent rLP2086 vaccine on 0- and 4-month schedule in primary study B1971012 and were followed up for 48 months during the stage 1 of this study.
- Stage 2, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 1-, and 6-month schedule in primary study B1971012 and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Stage 2, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0-, 2-, and 6-month schedule in primary study B1971010, B1971012 and B1971015 were included in this group. Only participants from B1971010 and B1971012 studies received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Stage 2, Group 4: rLP2086 (0-and 6-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0- and 6-month schedule in primary study B1971012 and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Stage 2, Group 5: rLP2086 (0- and 2-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0- and 2-month schedule in primary study B1971012 and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
- Stage 2, Group 6: rLP2086 (0- and 4-Month Schedule): Participants who received bivalent rLP2086 vaccine on 0- and 4-month schedule in primary study B1971012 and received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine at Visit 7 (approximately at Month 48) in booster stage of study B1971033.
Arm/Group | Stage1,Group 1:MCV4+Tdap+Saline (0-,2-,and 6-Month Schedule): | Stage 1, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule): | Stage 1, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule): | Stage 1, Group 4: rLP2086 (0-and 6-Month Schedule): | Stage 1, Group 5: rLP2086 (0- and 2-Month Schedule): | Stage 1,Group 6: rLP2086 (0- and 4-Month Schedule): | Stage 2, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) | Stage 2, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) | Stage 2, Group 4: rLP2086 (0-and 6-Month Schedule) | Stage 2, Group 5: rLP2086 (0- and 2-Month Schedule) | Stage 2, Group 6: rLP2086 (0- and 4-Month Schedule)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/101 | 0/277 | 0/116 | 0/86 | 0/46 | 0/59 | 0/92 | 0/64 | 0/54 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/59 | 1/92 | 2/64 | 1/54 | 0/32
Other Adverse Events (participants affected / at risk) | 4/70 | 0/101 | 1/277 | 0/116 | 2/86 | 1/46 | 56/59 | 90/92 | 62/64 | 53/54 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage1,Group 1:MCV4+Tdap+Saline (0-,2-,and 6-Month Schedule): (N=0) | Stage 1, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule): (N=0) | Stage 1, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule): (N=0) | Stage 1, Group 4: rLP2086 (0-and 6-Month Schedule): (N=0) | Stage 1, Group 5: rLP2086 (0- and 2-Month Schedule): (N=0) | Stage 1,Group 6: rLP2086 (0- and 4-Month Schedule): (N=0) | Stage 2, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) (N=59) | Stage 2, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) (N=92) | Stage 2, Group 4: rLP2086 (0-and 6-Month Schedule) (N=64) | Stage 2, Group 5: rLP2086 (0- and 2-Month Schedule) (N=54) | Stage 2, Group 6: rLP2086 (0- and 4-Month Schedule) (N=32)
Influenza like illness (General disorders) | NA | NA | NA | NA | NA | NA | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | NA | NA | NA | NA | NA | NA | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | NA | NA | NA | NA | NA | NA | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | NA | NA | NA | NA | NA | NA | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | NA | NA | NA | NA | NA | NA | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stage1,Group 1:MCV4+Tdap+Saline (0-,2-,and 6-Month Schedule): (N=70) | Stage 1, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule): (N=101) | Stage 1, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule): (N=277) | Stage 1, Group 4: rLP2086 (0-and 6-Month Schedule): (N=116) | Stage 1, Group 5: rLP2086 (0- and 2-Month Schedule): (N=86) | Stage 1,Group 6: rLP2086 (0- and 4-Month Schedule): (N=46) | Stage 2, Group 2: rLP2086 (0-, 1-, and 6-Month Schedule) (N=59) | Stage 2, Group 3: rLP2086 (0-, 2-, and 6-Month Schedule) (N=92) | Stage 2, Group 4: rLP2086 (0-and 6-Month Schedule) (N=64) | Stage 2, Group 5: rLP2086 (0- and 2-Month Schedule) (N=54) | Stage 2, Group 6: rLP2086 (0- and 4-Month Schedule) (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mite allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Genitourinary chlamydia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 5 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0/3
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1/3
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Borrelia test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 12 | 3 | 3 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 29 | 13 | 10 | 9
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 56 | 40 | 28 | 21
Injection site erythema (redness) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 19 | 13 | 15 | 2
Injection site pain (tenderness at injection site) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 54 | 86 | 57 | 48 | 27
Injection site swelling (swelling) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 19 | 11 | 8 | 3
Pyrexia (fever) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 15 | 9 | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 27 | 12 | 13 | 5
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 44 | 36 | 26 | 12
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT01543087/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT01543087/SAP_001.pdf